CLINICAL TRIAL: NCT04194112
Title: Diagnostic Performance and Predictive Capacity of Immediate Urine Cytology After Transurethral Resection of Non-Muscle Invasive Bladder Cancer; A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE 2398
Record Dates: First submitted 2019-12-07; First posted 2019-12-11 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMIBC patients (Other): Patients with primary or recurrent NMIBC for whom complete TURBT was done.
  Interventions: Diagnostic Test: immediate urine cytology

INTERVENTIONS:
Diagnostic Test: immediate urine cytology — Forty-eight hours after primary TURBT, IUC was retrieved and patients were scheduled for repeat TURBT 2 to 6 weeks later according to the predetermined protocol. The primary outcome was to determine the role of positive IUC to predict positive biopsy findings on repeat TURBT.

SUMMARY:
The current study aimed at prospectively assessing the performance of IUC as a predictive tool for residual tumor after primary TURBT of NMIBC, and possible future recurrence.

DETAILED DESCRIPTION:
The current study aimed at prospectively assessing the performance of IUC as a predictive tool for residual tumor after primary TURBT of NMIBC, and possible future recurrence.

ELIGIBILITY:
Inclusion Criteria:

-patients with primary or recurrent NMIBC for whom complete TURBT was done

Exclusion Criteria:

-Patients with concomitant CIS, upper tract urothelial tumors, biopsy proven muscle invasion, or low risk NMIBC (single, primary, Ta, G1 tumor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of IUC | It was assessed 48 hours after primary TURBT
  The primary outcome included assessment of the performance of IUC as a predictive tool for possible residual malignancy after primary TURBT. Thereafter, sensitivity (Sn), specificity (Sp), positive and negative predictive values (PPV, NPV) and overall accuracy of IUC as a preliminary step before repeat TURBT will be determined.

SECONDARY OUTCOMES:
The secondary outcome included the evaluation of predictive capacity of IUC for tumor recurrence in the study participants. | Within duration of follow up (4 years )
  The secondary outcome included the evaluation of predictive capacity of IUC for tumor recurrence in the study participants.

IPD SHARING:
Plan to Share IPD: Undecided